CLINICAL TRIAL: NCT06429163
Title: Impact of Pre-incisional Wound Infiltration and Hypogastric Plexus Block Using Ropivacaine on Postoperative Pain Following Laparoscopic Myomectomy: A Single-Center, Prospective, Randomized, Placebo-Controlled, Double-Blind Study
Brief Title: Pre-incisional Wound INfiltration and Hypogastric PLEXus Block Using Ropivacaine in Laparoscopic Myomectomy
Acronym: WINPLEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Nikita Kharlov, Head of Gynecology department, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WINPLEX
Record Dates: First submitted 2024-05-14; First posted 2024-05-24 (Actual); Results first posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Fibroid Uterus; Pain, Postoperative
Keywords: Uterine fibroid; Laparoscopic myomectomy; Postoperative pain; Pre-incisional infiltration; Hypogastric plexus block; EQ-5D questionnaire; Picker questionnaire; The Central Sensitization Inventory (CSI-R)
MeSH Terms: conditions — Leiomyoma; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: A single-centre prospective randomized placebo-controlled double-blind pilot study
Who Masked: Participant, Care Provider
Masking Description: All patients and clinicians involved in the study are unaware of the group assignment and syringe contents.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standart analgesia (Placebo Comparator): Standard postoperative analgesia (systemic non-steroidal anti-inflammatory drugs, paracetamol, opioid analgetics).
  Interventions: Procedure: Troacar site infiltration; Procedure: Superior hypogastric plexus block
- Troacar site infiltration (Active Comparator): Troacar site infiltration without SHP block
  Interventions: Procedure: Troacar site infiltration; Procedure: Superior hypogastric plexus block
- SHP block (Experimental): Standard systemic analgesia combined with troacar site infiltration and laparoscopic SHP block
  Interventions: Procedure: Troacar site infiltration; Procedure: Superior hypogastric plexus block

INTERVENTIONS:
Procedure: Troacar site infiltration — Infiltration of the anterior abdominal wall is performed with placebo or 0.2% ropivacaine diluted with physiological saline on a syringe in the volume of 20 ml - 5 ml for each incision. The drug is injected with a 22-gauge needle at a 90-degree angle.
Procedure: Superior hypogastric plexus block — At the beginning of the operation the camera is used to visualise the area of the promontorium. Next, a 1 mm laparoscopic puncture needle is inserted through a trocar in the suprapubic region and plunged into the upper part of the formed dome to a depth of no more than 1 cm. After positioning the needle retroperitoneally, an aspiration test is performed to prevent intravascular injection. Then, 20 ml of placebo or 0.2% ropivacaine diluted with physiological saline is slowly injected. At the end of the procedure, the retroperitoneal space swollen by the local anaesthetic is visualised in the promontorium.

SUMMARY:
The purpose of this study is to assess an impact of laparoscopic superior hypogastric plexus (SHP) block combined with preemptive troacar site infiltration on postoperative pain intensity following laparoscopic myomectomy.

DETAILED DESCRIPTION:
Patients randomized into 3 groups with a target ratio of 1:1:1 were included in the study: group 1 received standard systemic analgesia combined with troacar site infiltration and laparoscopic SHP block; group 2 received troacar site infiltration without SHP block; control group (group 3) received standard systemic analgesia alone. The primary endpoint was presented by assessing pain intensity using the numeric rating scale (NRS) at 4 hours postoperatively. Secondary endpoints included NRS dynamics at 2, 6, 8, 12, and 24 hours postoperatively, time to first mobilization, opioid use, and pain quality assessment.

ELIGIBILITY:
Inclusion Criteria

* Women aged ≥18 years.
* Indication for laparoscopic myomectomy due to ≥6 cm fibroid(s) or multiple fibroids.
* Ability to provide informed consent.

Exclusion Criteria

* FIGO type 7 subserosal pedunculated myoma.
* Conversion to laparotomy.
* Severe presacral adhesions preventing safe SHPB.
* Concomitant pelvic or abdominal surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- SHP Block: Standard systemic analgesia combined with troacar site infiltration and laparoscopic superior hypogastric plexus block
- Standart Analgesia (Control Group): Standard postoperative analgesia (systemic non-steroidal anti-inflammatory drugs, paracetamol, opioid analgetics).
Period: Overall Study
Arm/Group | SHP Block | Troacar Site Infiltration | Standart Analgesia (Control Group)
Started | 69 | 69 | 69
Completed | 66 | 65 | 67
Not Completed | 3 | 4 | 2
Not completed — uterine fibroid type 7 | 1 | 1 | 1
Not completed — severe adhesions | 1 | 2 | 1
Not completed — conversion to laparotomy | 0 | 1 | 0
Not completed — concomitant procedure | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SHP Block | Troacar Site Infiltration | Standart Analgesia | Total
Number analyzed (Participants) | 66 | 65 | 67 | 198
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 44.4 [39.1 to 46.9] | 44.1 [40.1 to 46.7] | 42.7 [38.9 to 44.8] | 43.4 [39.0 to 46.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 65 | 67 | 198
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Operative time, min [Median (Inter-Quartile Range); unit: min] — Although intraoperative parameters such as blood loss are measured during surgery rather than strictly before the intervention, they are not used as outcome measures in this study. These variables are collected to characterize the perioperative profile of the study cohorts and to confirm group comparability in terms of surgical complexity and intraoperative burden. In addition, intraoperative parameters are analyzed as potential risk factors for the development of significant postoperative pain, together with other baseline and perioperative characteristics.
  min | 97.5 [75 to 130] | 95 [68 to 120] | 95 [75 to 137.5] | 96 [75 to 117]
Blood loss, ml [Median (Inter-Quartile Range); unit: ml] — Although intraoperative parameters such as blood loss are measured during surgery rather than strictly before the intervention, they are not used as outcome measures in this study. These variables are collected to characterize the perioperative profile of the study cohorts and to confirm group comparability in terms of surgical complexity and intraoperative burden. In addition, intraoperative parameters are analyzed as potential risk factors for the development of significant postoperative pain, together with other baseline and perioperative characteristics.
  ml | 115 [50 to 200] | 100 [50 to 150] | 100 [50 to 200] | 105 [50 to 155]
Body mass index, kg/m^2 [Median (Inter-Quartile Range); unit: kg/m2] | 24.4 [21.9 to 28.4] | 25.1 [21.5 to 28.8] | 24.1 [20.9 to 27.6] | 24.5 [21.4 to 26.4]
Size of the largest myoma, mm [Median (Inter-Quartile Range); unit: mm] | 68 [55 to 80] | 69 [56 to 84] | 70 [62 to 80] | 69 [58 to 79]

OUTCOME MEASURES:

1. Primary Outcome: Pain Score
Description: Pain syndrome intensity 4 hours after laparoscopic myomectomy. The NRS (Numeric Rating Scale) score from 0-10 is a tool for self-reporting pain intensity, where 0 equals no pain and 10 equals the worst pain imaginable.
Time Frame: 4 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: NRS score (0-10 scale)
Arm/Group | SHP block | Troacar site infiltration | Standart analgesia (control group)
Number analyzed (Participants) | 66 | 65 | 67
NRS score (0-10 scale) | 2 [2.0 to 3.0] | 2 [2.0 to 4.0] | 4 [3.0 to 4.0]

2. Secondary Outcome: Pain Score Dynamics
Description: The NRS (Numeric Rating Scale) score from 0-10 is a tool for self-reporting pain intensity, where 0 equals no pain and 10 equals the worst pain imaginable.
Time Frame: 2, 6, 8, 12, and 24 hours postoperatively
Measure: Median (Inter-Quartile Range); unit: NRS score (0-10 scale)
Arm/Group | SHP block | Troacar site infiltration | Standart analgesia (control group)
Number analyzed (Participants) | 66 | 65 | 67
NRS score (0-10 scale)
  2 hours postoperatively | 2.5 [2.0 to 4.0] | 3.0 [2.0 to 4.0] | 4.0 [3.0 to 5.0]
  6 hours postoperatively | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 4.0]
  8 hours postoperatively | 2.0 [1.5 to 2.0] | 2.0 [2.0 to 3.0] | 2.0 [2.0 to 3.5]
  12 hours postoperatively | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 3.0]
  24 hours postoperatively | 2.0 [0.5 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 2.5]

3. Secondary Outcome: Mobilization
Description: Timing of post-surgery mobilization (hours after surgery)
Time Frame: Early postoperative period
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | SHP block | Troacar site infiltration | Standart analgesia (control group)
Number analyzed (Participants) | 66 | 65 | 67
Hours | 5.0 [4.0 to 7.0] | 7.0 [4.0 to 13.0] | 7.0 [5.0 to 11.5]

4. Secondary Outcome: Opioid Use
Description: Number of opioid administrations
Time Frame: Postoperative period, up to 48 hours
Measure: Number; unit: doses
Arm/Group | SHP block | Troacar site infiltration | Standart analgesia (control group)
Number analyzed (Participants) | 66 | 65 | 67
doses | 3 | 14 | 22

5. Secondary Outcome: Pain Localisation (Superficial/Deep)
Description: Patients were asked to characterize the predominant type of postoperative pain using a standardized questionnaire. Superficial pain was defined as somatic pain (localized, similar to muscle soreness), while deep pain was defined as visceral (diffuse, dull, similar to menstrual pain). Responses were used to evaluate the visceral pain component after surgery. Participants were allowed to report more than one type of postoperative pain.
Time Frame: Within 48 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | SHP block | Troacar site infiltration | Standart analgesia (control group)
Number analyzed (Participants) | 66 | 65 | 67
Participants
  Superficial pain | 30 | 15 | 21
  Deep (visceral) pain | 41 | 53 | 53

ADVERSE EVENTS:
Time Frame: Intraoperatively and within 48 after surgery
Description: Adverse events were prospectively monitored intraoperatively and during the first 48 hours after surgery. Serious adverse events were predefined as organ injury, bleeding requiring transfusion, reoperation, or unplanned intensive care unit admission. Non-serious adverse events included postoperative nausea and vomiting, urinary retention, and other perioperative complications. All adverse events were collected and categorized according to severity and reported in the Adverse Events tables.
Arm/Group | SHP Block | Troacar Site Infiltration | Standart Analgesia (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/65 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/65 | 0/67
Other Adverse Events (participants affected / at risk) | 0/66 | 0/65 | 0/67

LIMITATIONS AND CAVEATS:
Patient selection followed a per-protocol design rather than an intention-to-treat approach. This strategy was chosen deliberately, as the aim was not only to assess the efficacy and safety of the proposed technique, but also to refine its application during the surgical learning curve. Such a design ensured high group homogeneity and allowed evaluation of the method under optimal procedural conditions. However, it limited the generalizability of the findings to a broader patient population, par

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-12): https://cdn.clinicaltrials.gov/large-docs/63/NCT06429163/Prot_SAP_000.pdf